CLINICAL TRIAL: NCT07015372
Title: The Effect of Laughter Yoga on General Health Status, Perceived Stress Level, and Burnout in Psychiatric Nurses: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Stress, Burnout, and General Health in Psychiatric Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe DOST, Associate Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023_Dost_LaughterYoga
Record Dates: First submitted 2025-06-05; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Burnout; Perceived Stress; Occupational Stress; General Health; Psychiatric Nursing
Keywords: Laughter Yoga; Maslach Burnout Inventory; PSS-10; GHQ-28; Psychiatric Nurses; Nursing Interventions; Mental Health Promotion; Complementary Therapies; Burnout Prevention; Stress Reduction; Workplace Wellness
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two parallel groups: an experimental group receiving a structured laughter yoga program, and a control group receiving no intervention during the study period.
Masking Description: This is an open-label study. No parties were masked during the intervention or outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Laughter Yoga (Experimental): Participants in this group received a structured laughter yoga program consisting of 8 sessions over approximately four weeks. Each session lasted about 30 minutes and included clapping, breathing exercises, playful activities, and laughter exercises. Sessions were delivered face-to-face in small groups.
  Interventions: Behavioral: Laughter Yoga
- Control: No Intervention (No Intervention): Participants in this group did not receive any intervention during the study period. They continued their usual routines and duties. The same pre- and post-test assessments were applied as in the experimental group.

INTERVENTIONS:
Behavioral: Laughter Yoga — Laughter yoga intervention including clapping, breathing, childlike play, and laughter exercises, delivered in 8 sessions over 4 weeks to reduce stress and burnout and improve general health among psychiatric nurses.
  Arms: Experimental: Laughter Yoga

SUMMARY:
This study aims to examine the effects of laughter yoga on general health, perceived stress, and burnout among psychiatric nurses. Nurses working in psychiatric units are often exposed to high levels of occupational stress, which may impact their well-being and job performance. This trial was designed to evaluate the potential benefits of laughter yoga as a supportive intervention in this context.

DETAILED DESCRIPTION:
Psychiatric nurses frequently face emotionally intense situations, aggressive patient behaviors, and heavy workloads. These factors are known to contribute to elevated stress levels and burnout.

This study was conducted as a randomized controlled trial at a psychiatric hospital located on the Anatolian side of Istanbul, Türkiye. A total of 70 psychiatric nurses voluntarily participated and were randomly assigned to either an experimental group or a control group (n=35 per group).

The experimental group received an eight-session laughter yoga program, with each session lasting approximately 30 minutes. Sessions were held face-to-face in small groups and facilitated by a trained laughter yoga instructor. Each session included four components: warm-up and clapping exercises, deep breathing, childlike playfulness, and structured laughter activities. The control group received no intervention during the study period.

Data were collected before and after the intervention using the following validated tools:

Nurse Demographic Information Form

Maslach Burnout Inventory (MBI)

Perceived Stress Scale (PSS-10)

General Health Questionnaire (GHQ-28)

The study was approved by the relevant ethics committee, and all participants provided informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Being a psychiatric nurse at the specified hospital
* Volunteering to participate
* Not receiving psychiatric treatment currently

Exclusion Criteria:

* Chronic physical illnesses that could interfere
* Inability to attend all sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory (MBI) Total Score | Baseline and after 4 weeks (post-intervention)
  The Maslach Burnout Inventory (MBI) is used to assess burnout levels among psychiatric nurses. Scores range from low to high burnout. A decrease in score indicates reduced burnout. The scale has three subscales: emotional exhaustion, depersonalization, and personal accomplishment.
Change in Perceived Stress Level (PSS-10 Total Score) | Baseline and Week 4 (post-intervention)
  Perceived stress is measured using the 10-item Perceived Stress Scale (PSS-10). Total scores range from 0 to 40, with higher scores indicating greater perceived stress. A decrease in score reflects improvement.
Change in General Health Status (GHQ-28 Total Score) | Baseline and Week 4 (post-intervention)
  General health is evaluated using the General Health Questionnaire-28 (GHQ-28), which includes somatic symptoms, anxiety/insomnia, social dysfunction, and severe depression subscales. Total scores range from 0 to 28, with lower scores indicating better general health status.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe V Dost, Study Director — Bezmialem Vakıf Üniversitesi
Locations (1):
- Erenköy Ruh ve Sinir Hastalıkları Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset is currently being used for the preparation of a scientific publication. Data sharing may be considered after the publication process is complete, upon reasonable request and with appropriate approvals.